CLINICAL TRIAL: NCT05047315
Title: Evaluating a New Stool Based qPCR for Diagnosis of Tuberculosis in Children and People Living With HIV
Acronym: Stool4TB
Status: Active, not recruiting | Type: Observational
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Makerere University (Other); Amsterdam Institute for Global Health and Development (Other); Centro de Investigacao em Saude de Manhica (Other); Baylor Eswatini Clinical Centre of Excellence (COE) (Unknown); Research Center Borstel (Other); Fundação Manhiça (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: RIA2018D-2511
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Diagnoses Disease
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stool4TB aims to evaluate an innovative stool-based qPCR diagnostic platform (with the capacity to become a POC diagnostic tool) in the high TB and HIV burden settings of Mozambique, Eswatini and Uganda, under the hypothesis that it will narrow the extremely large TB case detection gap by improving TB confirmation rates in children and people living with HIV (PLHIV).

DETAILED DESCRIPTION:
Tuberculosis (TB) continues to be a leading cause of morbidity and mortality among children and people living with HIV (PLHIV). Despite significant progress in TB diagnostics, improvement of childhood TB diagnosis continues to be a major challenge and is a key pillar of the WHO "End TB Strategy". TB laboratory confirmation is particularly challenging in children and PLHIV given the difficulty in obtaining sputum samples, and the pauci-bacillary nature of disease. In consequence, bacteriological confirmation of pulmonary TB in young children and immunosuppressed PLHIV remains disappointingly low. Inability to bacteriologically confirm TB, results in both i) under diagnosis which leads to worse outcomes including increased mortality and ii) over or under diagnosis, and poor resource allocation. Given the limitations of currently available sputum-based diagnostic tests in these vulnerable populations, there is a need to develop new tools and identify easy to collect non-respiratory specimens which, combined, could improve bacteriological confirmation. Preliminary data suggest that a new platform, an innovative stool homogenization and DNA isolation method, adds value to existing sputum-based diagnostics by increasing the rates of bacteriological confirmation, and could also be useful as a monitoring tool for treatment response. This platform has the potential to be adapted to a point of care (POC) diagnostic and thus easily implemented in resource-constrained basic health care centres.

Objective: The aim of this project is to evaluate the diagnostic performance of the stool bead-based real-time quantitative PCR (qPCR) platform for TB diagnosis in children and PLHIV. This will be evaluated in the high TB and HIV burden settings of Mozambique, Eswatini and Uganda, under the hypothesis that it will narrow the large TB case detection gap by improving TB confirmation rates in children and PLHIV, while proving feasible and acceptable.

Primary objective:

• Evaluate the diagnostic accuracy of a stool-based real-time quantitative PCR for detecting DNA of Mycobacterium tuberculosis (MTB qPCR), compared to a composite reference standard (sputum and stool Xpert Ultra, sputum culture and urine TB-LAM).

Secondary objectives:

* Evaluate the diagnostic accuracy of the stool-based Mtb qPCR to individual sputum and stool Xpert Ultra, urine LAM, sputum smear and sputum culture (MGIT) results using a consensus clinical case definition as the reference standard.
* Evaluate the usefulness of the quantitative stool-based MTB qPCR platform as a tool to monitor treatment response for children and PLHIV.
* To create a biorepository of well characterized pediatric samples at each of the study sites to support the future development and evaluation of novel biomarker research.

Methodology: This is a prospective diagnostic evaluation study with a nested longitudinal cohort evaluation. During a 30-month recruitment period, people with presumptive TB will consecutively enroll being part of two study groups: Children less than 8 years of age, irrespective of HIV status (N=1295) and adults living with HIV, irrespective of immunological status (N=650). Sixty extra people will take part as healthy (asymptomatic) controls. After clinical, radiological and bacteriological evaluation, TB cases will be treated according to national guidelines. Participants diagnosed with TB will be followed up for 6 months since treatment initiation in order to assess treatment response and outcomes. A clinical case definition will be established as a reference standard and defined as any participant in whom a decision is made to start ATT (TB cases will be classified as confirmed or unconfirmed). Specifically, children will be classified into 3 distinct pediatric endpoint categories (confirmed TB, unconfirmed TB and Unlikely TB) based on bacteriological, radiological and clinical criteria, following international consensus guidelines.

ELIGIBILITY:
Inclusion Criteria:

Pediatric Cohort

* <8 years of age
* Identified with suspected PTB defined as follows:

  1. A child with ≥1 of the following criteria:

  <!-- -->

  1. Persistent unremitting cough (or cough significantly worse than usual in child with chronic lung disease including HIV-related) of >2 weeks duration, unresponsive to a course of appropriate antibiotics (when clinically indicated)
  2. Poor growth documented over the preceding 3 months [clear deviation from a previous growth trajectory and/or documented crossing of centile lines in the preceding 3 months and/or; weight-for-age, or weight-for-height Z-score of ≤2 in the absence of information on previous/recent growth trajectory AND not responding to nutritional rehabilitation (or to antiretroviral therapy if HIV-infected)]
  3. Persistent unexplained lethargy or reduced playfulness/activity reported by the caregiver.
  4. Persistent (>1w) unexplained fever (>38C), reported by a guardian or objectively recorded at least once;
  5. In infants 0-60 days, also: unresponsive neonatal pneumonia or unexplained hepatosplenomegaly OR sepsis-like illness (all other more common causes excluded and/or not responding to appropriate therapy/ broad-spectrum antibiotics/antivirals).

OR

2) Any duration of cough/ wheeze/ acute pneumonia with ≥1:

1. TB exposure. Either: i) Documented/Reported exposure to a known TB source case (regardless of smear status) in previous 12months OR ii) immunological evidence: positive IGRA or positive TST (defined as >5mm in HIV infected or severely malnourished, >10 otherwise)
2. Chest radiograph suggestive of TB.

Adult Cohort (WHO definition of a HIV-positive presumptive TB case)

* > 15 years of age
* Confirmed HIV infection (ELISA or molecular)
* Presenting at any health facility with any of the following: cough, fever, night sweats or unintentional weight loss (any duration).

Exclusion criteria

Participants will be excluded (both from study groups) if:

* Receiving TB treatment for >72 hours in previous 2 weeks
* History of TB treatment in the last year
* Refusal to provide consent for study participation or HIV testing when status is unknown
* Severe illness resulting in unstable condition
* Absolute contra-indication to any of sampling procedures required by the study (ie: acute severe asthma, pertussis syndrome etc.)

Ages: 0 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Our proposed diagnostic evaluation will be performed in three high TB/HIV burden settings in populations where the tests are intended to be used (presumptive adult pulmonary TB cases and presumptive intrathoracic pediatric TB cases). The study will enroll presumptive TB cases within two study groups:
  1. Children less than 8 years of age (irrespective of HIV status)
  2. Adults living with HIV (>15 years of age), irrespective of immunological status.
Sampling Method: Non-Probability Sample
Enrollment: 1945 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance qPCR test in stool samples | 2 months
  Diagnostic performance (Sensitivity, specificity, negative and positive predictive value) of the qPCR test in stool samples with respect to:
  1. bacteriologically confirmed tuberculosis as a composite gold standard of any of the other tests positive (including induced sputum and gastric aspirate Xpert Ultra and MGIT culture, stool Ultra or TB-LAM in urine)
  2. clinical reference standard case definition (S. Graham et al.; CID 2015).

SECONDARY OUTCOMES:
Comparison of diagnostic performance | 2 months
  Diagnostic performance of the qPCR test in stool compared to each of the other microbiological confirmation tests separately with respect to:
  A) bacteriologically confirmed tuberculosis as a composite excluding index/comparator).
  B) clinical l reference standard case definition (S. Graham et al.; CID 2015).
Monitor response to TB treatment | 6 months
  Ability of qPCR test in stool to monitor response to TB treatment, by comparing the change in readout over time while receiving TB treatment to that of Xpert Ultra in sputum and in stool.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto L García-Basteiro, MD, PhD, Principal Investigator — Barcelona Institute for Global Health; Elisa López Varela, MD, PhD, Study Director — Barcelona Institute for Global Health
Locations (3):
- Baylor Eswatini Clinical Centre of Excellence (COE), Mbabane, Eswatini
- Centro de investigação de Saúde de Manhiça, Manhiça, Maputo Province, Mozambique
- Makerere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kasule GW, Hermans S, Acacio S, Kay A, Nsubuga JK, Fernandez-Escobar C, Shiba N, Carratala-Castro L, Semugenze D, Mwachan P, Munguambe S, Ehrlich J, Lopez-Varela E, DiNardo AR, Cobelens F, Lange C, Joloba M, Mandalakas AM, Ssengooba W, Garcia-Basteiro AL; Stool4TB Global Partnership. Performance of stool Xpert MTB/RIF Ultra for detection of Mycobacterium tuberculosis among adults living with HIV: a multicentre, prospective diagnostic study. Lancet Microbe. 2025 Jul;6(7):101085. doi: 10.1016/j.lanmic.2025.101085. Epub 2025 Apr 4. PMID 40194533
- [Derived] Carratala-Castro L, Ssengooba W, Kay A, Acacio S, Ehrlich J, DiNardo AR, Shiba N, Nsubuga JK, Munguambe S, Saavedra-Cervera B, Manjate P, Mulengwa D, Sibandze B, Ziyane M, Kasule G, Mambuque E, Sekadde MP, Wobudeya E, Joloba ML, Heyckendorf J, Lange C, Hermans S, Mandalakas A, Garcia-Basteiro AL, Lopez-Varela E; Stool4TB Global Partnership. A stool based qPCR for the diagnosis of TB in children and people living with HIV in Uganda, Eswatini and Mozambique (Stool4TB): a protocol for a multicenter diagnostic evaluation. BMC Infect Dis. 2024 Feb 21;24(1):233. doi: 10.1186/s12879-023-08708-9. PMID 38383310